CLINICAL TRIAL: NCT04543136
Title: Exploratory Investigation on Performance and Safety of Newly Developed Intermittent Catheters in Male Users of Intermittent Catheters
Brief Title: Investigation of Non-CE Marked Intermittent Catheters.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CP323
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-08

CONDITIONS: Retention, Urinary
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent catheter; SpeediCath® Standard male (Active Comparator): Participants underwent two catheterizations with standard of care intermittent catheter: The first was performed by a trained nurse, the second by the participant later the same day.
  Interventions: Device: SpeediCath® Standard male
- New intermittent catheter Variant 1 for males (Experimental): Participants underwent two catheterizations with the new intermittent catheter Variant 1 for males: The first was performed by a trained nurse, the second by the participant later the same day.
  Interventions: Device: New intermittent Variant 1 catheter for males
- New intermittent catheter Variant 2 for males (Experimental): Participants underwent two catheterizations with the new intermittent catheter Variant 2 for males: The first was performed by a trained nurse, the second by the participant later the same day.
  Interventions: Device: New intermittent Variant 2 catheter for males

INTERVENTIONS:
Device: SpeediCath® Standard male — Intermittent catheterization through the urethra draining the bladder, using SpeediCath® Standard male.
  Arms: Intermittent catheter; SpeediCath® Standard male
Device: New intermittent Variant 1 catheter for males — Intermittent catheterization through the urethra draining the bladder, using the new Variant 1 catheter.
  Arms: New intermittent catheter Variant 1 for males
Device: New intermittent Variant 2 catheter for males — Intermittent catheterization through the urethra draining the bladder, using the new Variant 2 catheter.
  Arms: New intermittent catheter Variant 2 for males

SUMMARY:
Investigation of novel non-CE marked intermittent catheters. The study was a randomized, single blinded, cross-over investigation comparing two new catheters for males with a comparator catheter

DETAILED DESCRIPTION:
The CP323 study investigated a novel non-CE marked intermittent catheter, designed in two different variants, Variant 1 and Variant 2, respectively, and was conducted in Denmark. The study was a randomized, single blinded, cross-over investigation, comparing the two new variant catheters with a comparator catheter in 15 male IC users.

For each participant, the study thus contains three test visits/treatment arms (Comparator, Variant 1 and Variant 2, respectively), to which the 15 participants were randomized using a randomization sequence of six (i.e., there were six different random options for the order in which the participants tested the three catheters). There were 4-14 days between the test visits.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Minimum 18 years of age and with full legal capacity
* Daily intermittent catheterization for bladder management, with at least two catheters used on average pr. day, during the last 3 months
* Ability to self-catheterize
* Written informed consent, signed letter of authority and signed secrecy agreement given

Exclusion Criteria:

* Participation in any other clinical study during this investigation
* Symptoms of urinary tract infection as judged by the investigator
* Any know allergies towards ingredients in the products
* Relevant medical history that would prevent the subject from participation in the investigation (investigators judgement)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-03 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — Blegdamsvej 9, Urologisk klinik Afsnit 2112, Rigshospitalet, Denmark
Locations (1):
- Blegdamsvej 9, Urologisk klinik Afsnit 2112, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2020 and January 2021,16 users were recruited for the study from one site (Denmark) and encompassed the safety population.
Pre-assignment Details: The 16 recruited participant were randomized into the three treatment arms, using a randomization sequence of six. No participants were excluded, but two were discontinued at own wish after the baseline visit.
  Three participants had an adverse event; all were classified as mild, non-serious, two as 'Possibly related' and one as 'Unlikely related' (for details; see Adverse Events section).
  Thus, 14 participants constituted the intention to treat (ITT) population.
Groups:
- Comparator, Then Variant 2, Then Variant 1: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Comparator. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 1.
- Variant 2, Then Variant 1, Then Comparator: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Third intervention: Day of catheterization with Comparator.
- Comparator, Then Variant 1, Then Variant 2: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Comparator. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 2.
- Variant 1, Then Comparator, Then Variant 2: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Second intervention: Day of catheterization with Comparator. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 2.
- Variant 1, Then Variant 2, Then Comparator: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 1. Washout: 4-14 days. Second intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Third intervention: Day of catheterization with Comparator.
- Variant 2, Then Comparator, Then Variant 1: On three separate visits and in the listed random order, the participants underwent three interventions:
  First intervention: Day of catheterization with Variant 2. Washout: 4-14 days. Second intervention: Day of catheterization with Comparator. Washout: 4-14 days. Third intervention: Day of catheterization with Variant 1.
Period: Overall Study
Arm/Group | Comparator, Then Variant 2, Then Variant 1 | Variant 2, Then Variant 1, Then Comparator | Comparator, Then Variant 1, Then Variant 2 | Variant 1, Then Comparator, Then Variant 2 | Variant 1, Then Variant 2, Then Comparator | Variant 2, Then Comparator, Then Variant 1
Started | 3 | 3 | 2 | 3 | 2 | 3
Completed | 3 | 2 (Participant withdrew after baseline visit and prior to any interventions.) | 2 | 2 (Participant withdrew after baseline visit and prior to any interventions.) | 2 | 3
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population: Each treatment arm consisted of three test visits with 4-14 days between each crossover. On each visit, the participants underwent intermittent catheterization through the urethra, draining the bladder, and tested a different intermittent catheter: The comparator catheter (SpeediCath® Standard female), the new Variant 1 catheter, or the new Variant 2 catheter. For each visit and catheter tested, the participants underwent two catheterizations; the first catheterization was performed by a trained nurse and was followed by later same-day self-catheterization (i.e. performed by the participant).
Arm/Group | Total ITT Population
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 55 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 14
Number of participants with neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 9
Number of participants with non-neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 5
Number of participants in sitting catheterization position [Count of Participants; unit: Participants] | 8
Number of participants in standing catheterization position [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Residual Urine at 1st Flow-stop During Nurse Catheterization
Description: The residual urine at 1st flow-stop during nurse catheterization (i.e., catheterization performed by the nurse) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying/urination. This was assessed using a pressure sensor with time-logged weighing, meaning that a flow-stop was registered measuring the hydrostatic pressure at the outlet of an intermittent urinary catheter. Simultaneously, the collected urine was weighed and converted to volume, and the residual volume at first flow stop was calculated as the difference between the total urine volume collected and the volume collected at the first flow-stop.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: The intention to treat population (full analysis set) constituted all randomized subjects with a valid informed consent who was exposed to at least one product, and with valid information on at least one product with respect to the endpoints.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Intermittent Catheter; SpeediCath® Standard Male: Participants underwent intermittent catheterization through the urethra, draining the bladder. Two catheterizations were performed with standard of care intermittent catheter; SpeediCath® Standard male (active comparator). The catheterizations were performed by trained nurses followed by later same-day self-catheterization by the participants.
- New Intermittent Catheter Variant 1 for Males: Participants underwent intermittent catheterization through the urethra, draining the bladder. Two catheterizations were performed with new intermittent catheter Variant 1 for males. The catheterizations were performed by trained nurses followed by later same-day self-catheterization by the participants.
- New Intermittent Catheter Variant 2 for Males: Participants underwent intermittent catheterization through the urethra, draining the bladder. Two catheterizations were performed with new intermittent catheter Variant 2 for males. The catheterizations were performed by trained nurses followed by later same-day self-catheterization by the participants.
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
mL | 59.4 (99.6) | 13.1 (26.7) | 0.4 (1.66)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.074, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; Subject was included as a random effect, 'Visit' (Visit 1, 2 and 3) and 'Treatment' (comparator, Variant 1 and Variant 2) as fixed effects; Mean Difference (Final Values) = 45.0, 95% CI 2-sided [-4.5 to 94.5]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.022, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 58.8, 95% CI 2-sided [8.5 to 109.1]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.587, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-64.2 to 36.6]

2. Primary Outcome: Residual Urine at 1st Flow-stop During Self-catheterization
Description: The residual urine at 1st flow-stop during nurse catheterization (i.e., catheterization performed by the participant) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying/urination. This was assessed using a pressure sensor with time-logged weighing, meaning that a flow-stop was registered measuring the hydrostatic pressure at the outlet of an intermittent urinary catheter. Simultaneously, the collected urine was weighed and converted to volume, and the residual volume at first flow stop was calculated as the difference between the total urine volume collected and the volume collected at the first flow-stop.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
mL | 61.8 (117.7) | 5.7 (19.7) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.030, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 54.9, 95% CI 2-sided [5.3 to 104.4]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.015, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 61.8, 95% CI 2-sided [12.5 to 111.2]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.780, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-56.5 to 42.5]

3. Secondary Outcome: Post-void Residual Urine After Nurse Catheterization
Description: The volume of residual urine (urine left in the bladder) post catheterization (performed by the nurse) measured in triplicates using an ultrasound scanner.
Time Frame: Immediately after the procedure/catheterization, up to 15 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
mL | 24.6 (39.8) | 36.4 (56.5) | 12.7 (26.6)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.281, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.3, 95% CI 2-sided [-37.9 to 11.2]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.597, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [-18.3 to 31.7]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.116, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -20.0, 95% CI 2-sided [-45.1 to 5.0]

4. Secondary Outcome: Post-void Residual Urine After Self-catheterization
Description: The volume of residual urine (urine left in the bladder) post catheterization (performed by the participant) measured in triplicates using an ultrasound scanner.
Time Frame: Immediately after the procedure/catheterization, up to 15 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
mL | 33.9 (43.9) | 29.0 (53.16) | 27.0 (41.8)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.787, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-21.2 to 27.9]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.576, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-17.6 to 31.3]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.775, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-28.1 to 21.0]

5. Secondary Outcome: Insertion Discomfort During Nurse Catheterization
Description: Discomfort measured at catheter insertion (performed by nurse), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.59 (1.01) | 0.66 (1.16) | 1.20 (1.59)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.766, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.70 to 0.52]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.032, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.30 to -0.06]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.063, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.03 to 1.21]

6. Secondary Outcome: Urination Discomfort During Nurse Catheterization
Description: Discomfort measured during catheter urination/emptying (performed by nurse), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.44 (1.22) | 0.22 (0.33) | 0.17 (0.24)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.213, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.12 to 0.54]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.291, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.16 to 0.51]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.868, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.31 to 0.36]

7. Secondary Outcome: Withdrawal Discomfort During Nurse Catheterization
Description: Discomfort measured during catheter withdrawal (performed by nurse), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.41 (0.89) | 0.32 (0.44) | 0.59 (1.16)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.661, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.35 to 0.55]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.218, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.75 to 0.17]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.100, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.08 to 0.85]

8. Secondary Outcome: Overall Discomfort During Nurse Catheterization
Description: Discomfort measured for the entire catheterization procedure (performed by nurse), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.66 (1.68) | 0.79 (1.78) | 0.72 (1.09)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.701, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.80 to 0.54]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.438, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.96 to 0.42]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.689, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.55 to 0.83]

9. Secondary Outcome: Insertion Discomfort During Self-catheterization
Description: Discomfort measured at catheter insertion (performed by participant), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.24 (0.33) | 0.53 (0.73) | 0.73 (0.93)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.309, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.92 to 0.30]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.109, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.10 to 0.11]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.555, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.43 to 0.79]

10. Secondary Outcome: Urination Discomfort During Self-catheterization
Description: Discomfort measured during catheter urination/emptying (performed by participant), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.17 (0.26) | 0.18 (0.28) | 0.34 (0.59)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.896, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.35 to 0.31]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.320, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.49 to 0.16]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.390, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.19 to 0.47]

11. Secondary Outcome: Withdrawal Discomfort During Self-catheterization
Description: Discomfort measured during catheter withdrawal (performed by participant), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.15 (0.24) | 0.21 (0.31) | 0.55 (1.14)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.802, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.51 to 0.40]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.082, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.85 to 0.05]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.137, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.11 to 0.80]

12. Secondary Outcome: Overall Discomfort During Self-catheterization
Description: Discomfort measured for the entire catheterization procedure (performed by participant), using the Visual Analogue Scale (VAS). The VAS is a tool used to rate the intensity of certain sensations and feelings, e.g. discomfort/pain. It is a straight line of 10 cm (in this case horizontal) with one end meaning no discomfort/pain (0 cm) and the other end meaning the worst discomfort/pain imaginable (10 cm). The subject visualizes and marks a point on the line that matches the amount of discomfort/pain experienced. A high score reflects a worse outcome than a lower score.
Time Frame: Immediately after the procedure/catheterization, up to 5 min.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
Number analyzed (Participants) | 14 | 14 | 14
cm | 0.16 (0.24) | 0.38 (0.49) | 0.72 (1.25)
Statistical Analysis 1: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 1 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.525, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.89 to 0.46]
Statistical Analysis 2: Comparison: Intermittent Catheter; SpeediCath® Standard Male vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.098, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.24 to 0.11]
Statistical Analysis 3: Comparison: New Intermittent Catheter Variant 1 for Males vs New Intermittent Catheter Variant 2 for Males; Due to the exploratory nature of this investigation, no formal pass/fail criteria were applied; Test type: Superiority; p = 0.306, Mixed Models Analysis — The P-values were not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.33 to 1.02]

ADVERSE EVENTS:
Time Frame: Each participant was enrolled for 3 x 4-14 days for the entire investigation, thus a maximum of 42 days.
Description: The relationship to the investigational or comparator products was collected. The safety population constituted the subjects who had given informed consent and were thus 16 participants.
  An adverse event was reported as either: "Not related", "Unlikely related", "Possibly related", "Probably related", or "Definitely related", to the comparator to the Variant 1 or Variant 2 products.
Arm/Group | Intermittent Catheter; SpeediCath® Standard Male | New Intermittent Catheter Variant 1 for Males | New Intermittent Catheter Variant 2 for Males
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Catheter; SpeediCath® Standard Male (N=16) | New Intermittent Catheter Variant 1 for Males (N=16) | New Intermittent Catheter Variant 2 for Males (N=16)
Unlikely related (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Symptoms of urinary tract infection (UTI)
Possibly related (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Symptoms of urinary tract infection (UTI)
Possibly related (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Urinary tract infection (UTI)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT04543136/Prot_SAP_000.pdf